CLINICAL TRIAL: NCT02561390
Title: In-vivo Potency Evaluation of American Cockroach, Dog, Cat, Dust Mites and Mold Allergen Extracts Produced by Siriraj Hospital Comparing With Imported Extracts by Using Skin Prick Test.
Brief Title: Comparison Between spIgE and Skin Prick Test of Local and Imported Aeroallergens
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Principal Investigator, Nualanong Visitsunthorn, Prof, Mahidol University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Si521/2013
Record Dates: First submitted 2015-09-15; First posted 2015-09-28 (Estimated); Last update posted 2016-05-04 (Estimated); Status verified 2016-05

CONDITIONS: Immediate Hypersensitivity
MeSH Terms: conditions — Hypersensitivity, Immediate | interventions — Patch Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Skin prick test with aeroallergens (Experimental): Mean wheal diameters of SPT with commercial and local American coakroach, house dust mite, cat, dog and mold
  Interventions: Procedure: Skin prick test; Other: specific IgE measurement
- specific IgE measurement (Experimental): specific IgE levels of commercial and local American coakroach, house dust mite, cat, dog and mold
  Interventions: Procedure: Skin prick test; Other: specific IgE measurement

INTERVENTIONS:
Procedure: Skin prick test — skin prick test to American cockroach, dog, cat, dust mite and mold allergen extracts are performed
Other: specific IgE measurement — measure specific IgE of American cockroach, dog, cat, dust mite and mold

SUMMARY:
The prevalence of Allergic rhinitis(AR) and asthma was increased world wide. In 1998, ISAAC found that prevalence of AR and asthma inThailand was in moderately high group.

Tests for immediated reaction SPT and spIgE, were used for evaluated sensitization of allergen in patient. They guided the investigators for proper management as well as patient education. Clinician will use the result for choose allergen in case that might need immunotherapy.

SPT is safe and more economic for patient. Specific IgE has an advantage in patient who cannot withhold antihistamine prior SPT. In United state had a trial of result between SPT and spIgE for cockroach, cat, house dust mite and mold. It showed the correlation between two tests. In Thailand, the investigators haven't had data about it yet.

DETAILED DESCRIPTION:
SPT and specific IgE for allergens is necessary for allergen avoidance and specific immunotherapy. To have local allergen extracts will help the patients to easier get the appropriate management

ELIGIBILITY:
Inclusion Criteria:

* Patient with controlled Asthma and/or AR (mild to moderate severity) who were diagnosed in Allergy clinic and ENT clinic, Siriraj hospital
* SPT positve one of American Cockroach, House dust mite, cat, dog and mold.
* Patient were consented to trial.

Exclusion Criteria:

* Chronic disease such as heart disease, liver, renal and severe sepsis
* History of anaphylaxis
* Skin rash
* Pregnancy

Ages: 10 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 84 (Actual)
Dates: Start 2013-11; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
mean wheal diameter of SPT of local and imported allergen extracts and specific IgE levels | 18 months
  measure and compare SPT result of local and imported allergen extracts

CONTACTS AND LOCATIONS:
Overall Officials: Nualanong Visitsunthorn, Prof, Principal Investigator — Mahidol University
Locations (1):
- Faculty of Medicine Siriraj Hospital, Bangkoknoi, Bangkok, Thailand

REFERENCES:
- [Background] Worldwide variation in prevalence of symptoms of asthma, allergic rhinoconjunctivitis, and atopic eczema: ISAAC. The International Study of Asthma and Allergies in Childhood (ISAAC) Steering Committee. Lancet. 1998 Apr 25;351(9111):1225-32. PMID 9643741
- [Background] Vichyanond P, Jirapongsananuruk O, Visitsuntorn N, Tuchinda M. Prevalence of asthma, rhinitis and eczema in children from the Bangkok area using the ISAAC (International Study for Asthma and Allergy in Children) questionnaires. J Med Assoc Thai. 1998 Mar;81(3):175-84. PMID 9623008